CLINICAL TRIAL: NCT05737355
Title: Effect of ANKASCIN 568-P Products Regulating Blood Lipid- A Double-blind, Placebo-controlled Clinical Research
Brief Title: Effect of ANKASCIN 568-P Products Regulating Blood Lipid
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SunWay Biotech Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23 ANKASCIN 568-P
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This experiment adopts a block random assignment design, and the system assignment table (Block randomization, block size = 6) randomly generated by the program is given serial numbers and assigned to groups. The probability of assignment to each group is 1/2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANKASCIN 568-P Red yeast rice capsules (Experimental): ANKASCIN 568-P is a fermented product from the red yeast rice fungus <Monascus purpureus NTU 568>. It does not contain Monacolin K, an ingredient that may harm the human body, and is rich in new active ingredients. Take 2 red yeast rice capsules (each containing 440mg ANKASCIN 568-P) every day, and the control group takes 2 placebo capsules (containing equal weight maltodextrin) every day, respectively, at the 0th, 4th , , 12, 24, Collect blood samples for biochemical analysis and record the general body position measurement, blood pressure, blood lipid, blood sugar and other related changes of the subjects, and monitor the liver, kidney, and thyroid functions.
  Interventions: Dietary Supplement: ANKASCIN 568-P Red yeast rice capsules
- Placebo Capsules (Placebo Comparator): Maltodextrin was used as a placebo.
  Interventions: Dietary Supplement: Placebo Capsules

INTERVENTIONS:
Dietary Supplement: ANKASCIN 568-P Red yeast rice capsules — Product ingredients: ANKASCIN 568-P red yeast rice product 440 mg,microcrystalline ,cellulose,Maltodextrin; capsule shell composition: HPMC (hydroxypropyl methylcellulose), purified water, titanium dioxide, gellan gum.
  Arms: ANKASCIN 568-P Red yeast rice capsules
Dietary Supplement: Placebo Capsules — Maltodextrin was used as a placebo
  Arms: Placebo Capsules

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, parallel-controlled trial (24 weeks in total), divided into three periods (screening, treatment, and discontinuation follow-up)

DETAILED DESCRIPTION:
This study aims to investigate the effects of long-term consumption of red yeast rice products on blood lipid regulation and elevated high-density lipoprotein cholesterol (HDL-C), while also monitoring changes in the subjects' overall health. This randomized, double-blind, placebo-controlled trial aims to recruit 80 subjects, who will be randomly divided into two groups to receive either a red yeast rice product or a placebo for 24 weeks. The experimental group will take two red yeast rice capsules daily (each containing 440 mg of ANKASCIN 568-P), while the control group will take two similar-looking placebo capsules daily (containing an equal weight of maltodextrin). Blood samples will be collected and recorded for biochemical analysis at 0, 4, 12, and 24 weeks. General postural measurements will be taken, along with blood pressure, blood lipids, and blood glucose levels. Liver, kidney, and thyroid function will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female women over the age of 20 (women of childbearing age should not be pregnant or breastfeeding during the study period).
* A sane and communicative adult.
* 18≦BMI≦35.
* Sub-healthy people with simple dyslipidemia and those who have been judged by the doctor that they do not need to take hypolipidemic drugs for the time being, or those who insist on not taking drugs.
* Screening criteria Low-density lipoprotein cholesterol (LDL-C): 130~190 mg/dL. screening criteria and high-density lipoprotein cholesterol (HLDL-C): below 50 mg/dL.
* Those without other serious diseases (cancer, heart failure, diabetes, myocardial infarction, liver cirrhosis, moderate to severe liver and kidney dysfunction, stroke, etc.).
* During the experiment, the daily routine and eating habits should be maintained and not changed deliberately.

Exclusion Criteria:

* Triglyceride TG≧500 mg/dL.
* Blood pressure value: systolic blood pressure ≧ 200 mmHg or diastolic blood pressure ≧ 140 mmHg.
* Patients with moderate or severe abnormal liver and kidney function (generally referring to serum aminopyruvate converting enzyme (SGPT), serum glutamate phenylacetate transaminase (SGOT) are more than 3 times the upper limit of normal or have been diagnosed Liver cirrhosis, or glomerular filtration rate eGFR≦30 ml/min/1.73m2).
* Pregnant or lactating women.
* Those who take traditional Chinese medicine mainly based on red yeast rice.
* Those who have undergone surgery within one month.
* Those who have serious diseases such as heart, liver, kidney, and hematopoietic system, mentally ill patients who do not meet the inclusion criteria, fail to use the test product according to the regulations so that the efficacy or safety cannot be judged due to incomplete data.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Improves total cholesterol (TC) | 24 weeks
  Compare the improvement of total cholesterol (TC) between the test group and the placebo group after taking red yeast rice capsules or placebo capsules for 24 weeks. According to the results of Section 9. Statistical method, whether there is a statistical difference between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: WEN-HUI FANG, Ph. D., Principal Investigator — Chief of Family medicine department
Locations (1):
- Tri-Service General Hospital, National Defense Medical Center, Taipei city,, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hajar R. Risk Factors for Coronary Artery Disease: Historical Perspectives. Heart Views. 2017 Jul-Sep;18(3):109-114. doi: 10.4103/HEARTVIEWS.HEARTVIEWS_106_17. No abstract available. PMID 29184622
- [Result] Lin YL, Wang TH, Lee MH, Su NW. Biologically active components and nutraceuticals in the Monascus-fermented rice: a review. Appl Microbiol Biotechnol. 2008 Jan;77(5):965-73. doi: 10.1007/s00253-007-1256-6. Epub 2007 Nov 22. PMID 18038131
- [Result] Echaniz-Laguna A, Mohr M, Tranchant C. Neuromuscular symptoms and elevated creatine kinase after statin withdrawal. N Engl J Med. 2010 Feb 11;362(6):564-5. doi: 10.1056/NEJMc0908215. No abstract available. PMID 20147729
- [Result] Hsu LC, Hsu YW, Hong CC, Pan TM. Safety and mutagenicity evaluation of red mold dioscorea fermented from Monascus purpureus NTU 568. Food Chem Toxicol. 2014 May;67:161-8. doi: 10.1016/j.fct.2014.02.033. Epub 2014 Feb 28. PMID 24582683
- [Result] Lee CL, Wen JY, Hsu YW, Pan TM. Monascus-fermented yellow pigments monascin and ankaflavin showed antiobesity effect via the suppression of differentiation and lipogenesis in obese rats fed a high-fat diet. J Agric Food Chem. 2013 Feb 20;61(7):1493-500. doi: 10.1021/jf304015z. Epub 2013 Feb 8. PMID 23360447
- [Result] Lee CL, Kung YH, Wu CL, Hsu YW, Pan TM. Monascin and ankaflavin act as novel hypolipidemic and high-density lipoprotein cholesterol-raising agents in red mold dioscorea. J Agric Food Chem. 2010 Aug 25;58(16):9013-9. doi: 10.1021/jf101982v. Epub 2010 Jul 28. PMID 20666456
- [Result] Lee CL, Hung YP, Hsu YW, Pan TM. Monascin and ankaflavin have more anti-atherosclerosis effect and less side effect involving increasing creatinine phosphokinase activity than monacolin K under the same dosages. J Agric Food Chem. 2013 Jan 9;61(1):143-50. doi: 10.1021/jf304346r. Epub 2012 Dec 24. PMID 23237237
- [Result] Chen CL, Pan TM. Red mold dioscorea: a potentially safe traditional function food for the treatment of hyperlipidemia. Food Chem. 2012 Sep 15;134(2):1074-80. doi: 10.1016/j.foodchem.2012.03.019. Epub 2012 Mar 16. PMID 23107730
- [Result] Lee CL, Wen JY, Hsu YW, Pan TM. The blood lipid regulation of Monascus-produced monascin and ankaflavin via the suppression of low-density lipoprotein cholesterol assembly and stimulation of apolipoprotein A1 expression in the liver. J Microbiol Immunol Infect. 2018 Feb;51(1):27-37. doi: 10.1016/j.jmii.2016.06.003. Epub 2016 Jun 24. PMID 27422746
- [Result] Liu SF, Wang YR, Shen YC, Chen CL, Huang CN, Pan TM, Wang CK. A randomized, double-blind clinical study of the effects of Ankascin 568 plus on blood lipid regulation. J Food Drug Anal. 2018 Jan;26(1):393-400. doi: 10.1016/j.jfda.2017.04.006. Epub 2017 Jun 1. PMID 29389579